CLINICAL TRIAL: NCT01642264
Title: Web-Based Respiratory Education About Tobacco and Health (WeBREATHe) Phase II
Brief Title: Web-Based Respiratory Education About Tobacco and Health Phase II
Acronym: WeBREATHe II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HL083540
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Intervention (Training) Condition; Control (Delayed Training) Condition
Keywords: Tobacco Cessation; Continuing Education; Pediatric; Respiratory Therapist; Nurse
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Delayed Training) Condition (No Intervention): Participants in this condition were assessed at 1 week, 1 month and 3 months post-enrollment, and were provided access to the WeBREATHe training website upon completion of their 3-month assessment.
- Intervention (Training) Condition (Experimental): In this condition, participants used the WeBREATHe training program website for 1 week, and completed assessments at 1 week, 1 month, and 3 months post-training.
  Interventions: Behavioral: WeBREATHe Training Program

INTERVENTIONS:
Behavioral: WeBREATHe Training Program — The WeBREATHe Training Program is a web-based, interactive training program to teach pediatric respiratory therapists, nurses and nurse practitioners how to help their patients' parents to quit smoking.
  Arms: Intervention (Training) Condition

SUMMARY:
The primary aim of this study was to develop an interactive Internet-based program (WeBREATHe: Web-Based Respiratory Education About Tobacco and Health) to train pediatric respiratory therapists and nurses to provide brief, hospital-based tobacco cessation interventions to parents of pediatric patients. The WeBREATHe program was based on a Phase I prototype which was evaluated with 50 pediatric respiratory therapists and nurses.

In Phase II, the investigators redesigned and expanded the program with input from 50 educators, nurses and respiratory therapists from Cincinnati Children's Hospital Medical Center. Then the investigators evaluated the Phase II program in a randomized trial in which 215 respiratory therapists and nurses from two large, urban children's hospitals were randomly assigned within hospital to either the Intervention (Training) Condition, or to a Delayed Treatment (Training) Control condition.

Participants' demographic and tobacco use history were measured at baseline, and tobacco cessation intervention behaviors, attitudes, knowledge, perceived barriers, and self-efficacy regarding delivery of a tobacco cessation intervention were measured at baseline, 1 week post-training, and at 3 months post-training. User satisfaction measures were also collected at 1 week post-training from Intervention Condition participants. The investigators hypothesized that participants in the Intervention Condition would have increased tobacco cessation behaviors, positive attitudes and self-efficacy, and decreased perceived barriers than participants i the Delayed-Treatment Control Condition.

Following evaluation, the investigators developed a final version of the interactive training program and created the administrative infrastructure for a marketable product.

ELIGIBILITY:
Inclusion Criteria:

* Must be a respiratory Therapist, nurse or nurse practitioner at the 2 pediatric hospitals participating in the study.
* Must be at least 18 years of age.

Exclusion Criteria:

* Under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Performance of Ask, Advise, Assess, Assist and Arrange Behaviors | 3 months post-enrollment
  14 items measured on a 5-point Likert scale of frequency. Ask = asking all patients' parents about tobacco use and documenting use in the patients' charts.
  Advise = discussing health hazards of tobacco use and giving direct advice to quit.
  Assess = determining parents' level of readiness to quit. Assist = discussing strategies or techniques to quit, setting a specific date to quit, discussing pharmacotherapy for tobacco cessation, giving written self-help materials to tobacco users.
  Arrange = discussing local tobacco cessation resources and making a referral to a tobacco quit line.

SECONDARY OUTCOMES:
Attitudes towards provision of tobacco cessation interventions | 3 months post-enrollment
  9 items. Level of agreement measured on a 5-point Likert scale on 9 statements measuring attitudes towards provision of tobacco cessation interventions to patients' parents in pediatric settings. For example, "It is appropriate for pediatric RTs and RNs to assess and document their patients' exposure to secondhand smoke (e.g., family members' tobacco use)."
Perceived Barriers | 3 months post-enrollment
  7 items measured on a 5-point Likert scale. Participants rate the level of routine barriers to provision of tobacco cessation interventions in pediatric settings, (e.g., lack of training, lack of time, lack of resources).
Self-Efficacy | 3 months post-enrollment
  6 items measured on a 5-point Likert scale. Participants rate their agreement to statements of perceived self-efficacy to perform Ask, Advise, Assess, Assist and Arrange behaviors (e.g., "I can ask my patients' parents about their smoking.")